CLINICAL TRIAL: NCT06172179
Title: Construction and Validation of a Risk Prediction Model for Secondary Vertebral Fracture in Patients With Osteoporotic Vertebral Compression Fractures After Percutaneous Vertebroplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-1155-01
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Osteoporotic Vertebral Fracture; Prediction Model

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Sun Yat-sen memorial hospital
  Interventions: Other: No interventions
- Second People's Hospital of Foshan City
  Interventions: Other: No interventions
- The Fifth People's Hospital of Nanhai District, Foshan City
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — All procedures are observation. No intervention in this study.

SUMMARY:
"Retrospectively collecting clinical data from post-PVA (Percutaneous Vertebroplasty) patients, recording incidences of secondary vertebral fractures, and conducting statistical analysis to create a risk prediction model for recurrent fractures."

ELIGIBILITY:
Inclusion Criteria:

1. Meets the diagnostic criteria for primary osteoporosis as per the Osteoporosis Diagnosis and Treatment Guidelines (2022);
2. No history of high-energy trauma;
3. Patient complains of pain in the lumbar region, confirmed by MRI showing a newly developed vertebral fracture from T5 to L5 (i.e., MRI shows low signal on T1 and high or slightly high signal on T2);
4. Has undergone Percutaneous Vertebroplasty (PVA) treatment.

Exclusion Criteria:

1. Incomplete imaging or medical record data;
2. History of spinal surgeries other than PVA;
3. Pre-existing symptoms of spinal cord compression or nerve root injury;
4. Patients undergoing PVA treatment due to conditions such as tumors, vascular malformations, infections, or symptomatic Schmorl's nodes;
5. Chronic conditions like Kummell's disease or non-union of old fractures;
6. Concurrent vertebral burst fractures;
7. Diagnosis of central nervous system diseases such as dementia or stroke before or during the follow-up period post-PVA procedure;
8. History of violent trauma after PVA procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Older population with osteoporosis, who have undergone vertebral augmentation procedures due to osteoporotic vertebral fractures.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
secondary vertebral fractures | 2 years post-operative
  Recording the secondary vertebral fractures

CONTACTS AND LOCATIONS:
Overall Officials: Chunhai Li, MD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen memorial hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No